CLINICAL TRIAL: NCT06708039
Title: Self-Management and Exercise Programme Using Mobile Instant Messaging Application for Older Adults Living with Chronic Knee Pain.
Acronym: SMEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Responsible Party: Principal Investigator, Suliza binti Sulaiman, Principal Investigator, International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IREC 2024-226
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Chronic Knee Pain
Keywords: Self-management; Exercise; WhatsApp; Older Adults; Chronic Knee Pain
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The experimental group will receive the self-management and exercise programme, which will be delivered using mobile messaging application (WhatsApp), twice per week for five weeks. In addition, the experimental group will also continue their Elderly Day Care Centre routine activities. On the other hand, the control group will continue their Elderly Day Care Centre routine activities only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Instant Messaging Application based Self-Management and Exercise Programme (SMEP) (Experimental): The experimental group will receive the self-management and exercise programme, which will be delivered using mobile messaging application (WhatsApp), twice per week for five weeks. In addition, the experimental group will also continue their Elderly Day Care Centre routine activities.
  Interventions: Other: Mobile Instant Messaging Application based Self-management and Exercise Programme (SMEP)for Older Adults with Chronic Knee Pain.
- Control Group (No Intervention): The control group will continue their PAWE routine activities only

INTERVENTIONS:
Other: Mobile Instant Messaging Application based Self-management and Exercise Programme (SMEP)for Older Adults with Chronic Knee Pain. — The Mobile Instant Messaging Application based self-management and exercise programme (SMEP) consists of 10 short videos of self-management on chronic knee pain in older adults (5-10 minutes/video), 10 short videos of exercise interventions (5-10 minutes/video) and group discussions (10-20 minutes/session) with each video/session focusing on different content. A WhatsApp group that includes all participants in the intervention group will be created to deliver the three components of the program twice a week for five weeks. At the end of each session, they will be given the power point slides from the self-management video in Pdf format and an e-pamphlet of the exercise video. A total of 30-40 minutes will be allocated for each session to allow for socialization between the participants and researcher and also for a question and answer session.
  Arms: Mobile Instant Messaging Application based Self-Management and Exercise Programme (SMEP)

SUMMARY:
The goal of this Cluster Randomised, controlled trial (CRT, with two parallel groups pre- and post-test design) is to evaluate the potential effects of the self-management and exercise programme (SMEP) for older adults living with chronic knee pain which is delivered using mobile instant messaging application. The main questions it aims to answer are:

1. Are there any change in pain, physical function, mental well-being, the risk of fall, health belief and self-efficacy and quality of life after the intervention is carried out at week 5?
2. Are there any significance difference in pain, physical function, mental well-being, the risk of fall, health belief and self-efficacy and quality of life between the experimental and control group at baseline and week 5.
3. What are the factors related to the adherence to programme within 5 weeks it is delivered.
4. What are the factors that facilitates or inhibits the implementation process of the programme

Selected clusters will be randomized into either experimental or control group. The experimental group will receive the self-management and exercise programme, which will be delivered using mobile messaging application, twice per week for five weeks. In addition, the experimental group will also continue their Elderly Day Care Centre routine activities. On the other hand, the control group will continue their Elderly Day Care Centre routine activities only

DETAILED DESCRIPTION:
3.1 Study Type and Design A cluster randomized controlled trial (CRT) with two parallel groups (experimental vs control) pre- and post-test design will be utilized to conduct this study. Four clusters of Elderly Day Care Centre will participate in this study, where each two will be randomized into either experimental or control group by using a computer generated table of random numbers by a person external to the study. The experimental group will receive WhatsApp-based self-management and exercise programme (SMEP) twice per week for five weeks in addition to Elderly Day Care Centre routine activities that they normally receive. On the other hand, the control group will continue the routine activities only. The routine activities in Elderly Day Care Centre include the medical care (pharmacological and non-pharmacological treatment) prescribed by their healthcare professionals, various programmes (E.g. religion, recreation, therapy, rehabilitation and health talk programme) and appropriate training or courses.

At first appointment, both groups will receive an educational session by the researcher that explain briefly about the programme, anatomical of the knee, chronic knee pain, risk factors of knee pain, management of knee pain, self-management and exercise as a treatment, recommended exercise and pain management techniques in a two-hour educational session. In addition to the first educational session at the Elderly Day Care Centre, participants in the intervention group will receive all the self-management and exercise content through the mobile instant messaging application (WhatsApp). However, participants allocated to the control group will be given the component of the programme after finishing the study (after 5 weeks).

The researcher will only meet the participants once at the beginning of the study. Data on demographics, clinical, Knee Pain Scoring Tools (KNEST) and Physical Activity Readiness Questionnaire for Everyone (PAR-Q) will be collected directly from the participants from both groups at the beginning of the study. All outcome measures will be measure before the initiation of the program (baseline), and then measured again at five weeks of training (post-training). Questionnaires in Malay will be used to measure pain, physical function, mental well-being, the risk of fall, health belief and self-efficacy and quality of life.

The SMEP will be develop by findings from the systematic literature reviews and relevant evidence based including theory that support choices for the intervention content. The development of the programme will be guided by the UK MRC framework. The programme were developed and adopted based on previous studies that had showed the significance effect of that particular programme . However, this programme is more focusing on the management of chronic knee pain for older people.

This programme consists of 10 short videos of self-management on chronic knee pain in elderly (5-10 minutes/video), 10 short videos of exercise interventions (5-10 minutes/video) and group discussions (10-20 minutes/session) with each video/session focusing on different content.

A WhatsApp group that includes all participants in the intervention group will be created to deliver the three components of the program twice a week for five weeks. At the end of each session, they will be given the power point slides from the self-management video in Pdf format and an e-pamphlet of the exercise video. A total of 30-40 minutes will be allocated for each session to allow for socialization between the participants and researcher and also for a question and answer session. The programme will be carried out at a particular time of day, though the participants will open the messages at their convenient time. Reminders will be sent out to participants on the WhatsApp group at 10pm before the day the programme will be carried out, and by 8am on the actual day of the programme. The viewer info in WhatsApp will be used to assess if the contents of the programme are successfully delivered. Participants will be allowed to seek for advice or ask any questions at any time during the programme.

In addition, both the intervention and control groups will receive an activity diary to track their progress and symptoms, in the form of a Google form on their WhatsApp groups (Control group will have a separate Whatsapp group). Participants in the intervention group must fill out their diary twice a week for five weeks, while those in the control group will log their activities weekly from the start to the fifth week. If both groups of participants do not submit their activity diary before the next intervention session, they will receive individual WhatsApp messages to remind them to follow the prescribed intervention (for intervention group only) and submit the diary (for both groups).

3.2 Study Population This study will be conducted at four clusters of Elderly Day Care Centre from 12th to 31st November 2024. The study population will be all older adults with chronic knee pain attending these clusters during the study period. An older adult in this study is defined as those aged 60 years and above. The chronic knee pain is based on the older adults' self-report of having the pain for more than 3 months. Those who meet the study criteria listed in Section 3.3 and 3.4 will be selected to be included in this study using the random sampling method.

3.3 Inclusion Criteria i. Able to meet programme requirement - screening via KNEST and PAR-Q. ii. Owning a smartphone, tablet, or computer with an internet connection and WhatsApp application; and being able to use the device without assistance.

iii. Independently mobile either with or without a walking aid. iv. Able to communicate in Malay. v. Able to read and write in Malay.

3.4 Exclusion Criteria

i. Knee replacement / lower limb arthroplasty. ii. Intraarticular injections within the past six months. iii. Significant musculoskeletal issues (e.g. inflammatory arthritis, connective tissue diseases, fibromyalgia, severe osteoporosis, peripheral neuropathy, or gout).

iv. Unstable medical or psychiatric conditions. v. Severe cognitive, auditory or visual impairment.

3.5 Withdrawal Criteria Involvement in this study is voluntary. The participant has the right to discontinue (withdraw) from the study at any time and level, without compromising their present and future Elderly Day Care Centre daily routine activities.

3.6 Sample Size Calculation of the sample size for this study will be based on the conservative estimation of a clinically meaningful improvement, which was considered to be 15% of the baseline value. The recommendation for the sample size of the participants is between 34 and 116 for each groups (α = 0.05, power = 0.80) by using the effect size of the outcomes as at week 12 (0.44-0.75). A sample size of 68 participants will be required with 34 subjects for each group to estimate expected differences in the level of pain for the intervention and control groups. By allowing for 20% withdrawal by 12 weeks, estimation of 82 participants in both groups (41 each) will be recruiting from the four (4) Elderly Day Care Centre for the desired power of 80% and significance of 0.05 (2-tailed) for the analyses.

3.7 Study Duration and Timeline The study will start on 1 June 2024 and end on 31 January 2025.

* Stage 1: Modelling process and outcomes - 5 months
* Stage 2: Data collection and data analysis - 3 months
* Stage 3: Presentation and publication - 5-6 months The duration of the participant's involvement is 3 months starting from the middle of November 2024 and ending in January 2025.

3.8 Statistical Analysis Plan

Data analysis in this study will be carried out using Statistical Package for the Social Sciences (SPSS) Version 23. Descriptive statistics will be used to summarise participants' demographic characteristics and clinical information. These include frequencies and percentages for categorical variables and means and standard deviations (SD) for continuous variables. The demographic characteristics will be compared between the intervention group and control group by using Chi-square test for categorical data and independent t-test or Mann-Whitney U test for continuous data that are normally and non-normally distributed respectively. Independent t-test or Mann-Whitney U test will also be used to compare outcomes between both groups. Depending on the normality of data, Measures Analysis of Variance (RMANOVA) or Friedman test will be employed to examine the changes in the outcomes from baseline to week 5 for the intervention group. A p-value <0.05 is considered statistically significant.

3.9 Risk and benefit to study participants As identified through literature review, there are no serious side effects known to be caused by this study. Participants are requiring to read and sign written consent to participate in this study, which may cause some discomfort. The data collection process involves the active involvement of the participants to perform some exercise and do self-management which may also cause some discomfort. All participants will continue routine activities in Elderly Day Care Centre. The experimental group will receive an additional programme that is SMEP, which involves some physical and psychosocial risk to the subject.

The risk for participants receiving the research intervention is minimal because the exercise schedule given is of low to moderate intensity. However, the risk may be due to existing related diseases among the elderly. Potential side effects for seniors who exercise include the potential for chest pain, muscle pain, dizziness, nausea, vomiting, extreme fatigue, discomfort and difficulty. Participants are allowed to stop exercising at any time if they feel uncomfortable.

In terms of benefits, participants may get the benefits from this programme. All the information obtained from this research will be able to help in improving treatment methods or management of suffering patients from chronic knee pain. The results of this study are expected to provide implications for the daily treatment of elderly people suffering from chronic knee pain and if this method is found to be effective; can improve a better understanding of knee pain management; reduce pain or discomfort in the knee; and then be able to optimize the ability of physical activity, daily activities, mental well-being which in turn leads to a better quality of life.

3.10 Risk Benefit Assessment As stated above, there is minimal risk from this study. Study findings shall potentially greatly improve treatment outcomes. The expected benefit outweighs the minimal risk to subjects and thus this study should be supported. If any injuries do occur as a direct result of participating in the study, treatment for such injuries shall be provided or paid for by the researcher. However, the researchers will not be responsible for medical expenses for diseases or treatments that existed before their participation in this research. However, participants still do not lose any of their legal rights to compensation even if they have signed this form.

3.11 Ethics of Study The study will be conducted according to the ethical principles listed in the Declaration of Helsinki and Malaysian Good Clinical Practice Guideline. There will be no potentially vulnerable participants involved in this study as older adults with unstable medical or psychiatric conditions or severe cognitive, auditory or visual impairment are excluded from the study. This study also had been approved by International Islamic University Malaysia (IIUM) Research Ethics Committee (IREC) with ID Num. REC 2024-226 and registration approved by Malaysian National Medical Research Register with NMRR ID-24-01930-IDO

3.12 Informed Consent/Assent Process Participants shall be informed of the study during their usual visit to Elderly Day Care Centre. They will be requested to contact investigators if they are interested. An appointment will be made where the patient information sheet will be provided and explained to them. If they are willing to participate, the consent forms will be signed and dated. If they need to, they are allowed to take the information sheet home to consult with their family members, and another day for getting consent arranged.

3.13 Privacy and Confidentiality Subject's names will be kept on a password-protected database and will be linked only with a study identification number for this research. The identification number instead of patient identifiers will be used on subject data sheets. All data will be entered into a computer that is password-protected. On completion of study, data in the computer will be copied to CDs and the data in the computer erased. CDs and any hardcopy data will be stored in a locked office of the investigators and maintained for a minimum of three years after the completion of the study. The CDs and data will be destroyed after that period of storage. Participants will not be allowed to view their personal study data, as the data will be consolidated into a database. Participants can write to the investigators to request access to study findings

3.14 Conflict of Interest The investigators declare they have no conflict of interest.

3.15 Publication Policy No personal information will be disclosed and participants will not be identified when the findings of the study are published.

3.16 Termination of Study The researcher may decide to terminate the study at any time. Participants will be informed if the study is terminated and follow-up visits will be arranged if needed.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of having the pain for more than 6 months.
* Able to meet programme requirement - screening via KNEST and PAR-Q.
* Owning a smartphone, tablet, or computer with an internet connection and WhatsApp application; and being able to use the device without assistance.
* Independently mobile either with or without a walking aid.
* Able to communicate in Malay.
* Able to read and write in Malay.

Exclusion Criteria:

* Knee replacement / lower limb arthroplasty.
* Intraarticular injections within the past six months.
* Significant musculoskeletal issues (e.g. inflammatory arthritis, connective tissue diseases, fibromyalgia, severe osteoporosis, peripheral neuropathy, or gout).
* Unstable medical or psychiatric conditions.
* Severe cognitive, auditory or visual impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain Trough Knee Injury and Osteoarthritis Outcome Score subscales of pain (KOOS-pain) at 5 weeks. | From enrollment to the end of treatment at 5 weeks
  KOOS-pain - Included nine questions about pain that score on a Likert scale with five answer alternatives ranging from 0 (no problem) to 4 (extreme problem). Each of the five scores is calculate as the sum of the items and scores between 0 and 100 represent the percentage of total possible score achieve. Zero representing extreme knee problems and 100 representing no knee problems
Change from Baseline in the Physical Function Trough Knee Injury and Osteoarthritis Outcome Score (KOOS) subscales of symptoms (KOOS-symptoms), function in daily living (KOOS-ADL), function in sports and recreation (KOOS-sport/rec) at 5 weeks. | From enrollment to the end of treatment at 5 weeks
  Another three (3) subscale in KOOS that provide information about the disability impact from knee injury and associated problems on recreational activities and at the same time also it provides a good indicator for physical performance. All items in each subscale contain questions that were scored on a Likert scale of 0 (no problem) to 4 (extreme problem), where subscale symptoms (7 items); ADL Function (17 items); Sport and Recreation Function (5 items). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Change from Baseline in Mental Well-being Trough Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) at 5 weeks. | From enrollment to the end of treatment at 5 weeks
  SWEMWBS is a short version of the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) and enable to monitor of mental wellbeing in the general population that is widely used globally. It uses seven of the WEMWBS's 14 statements about thoughts and feelings, which relate more to functioning than feelings and so offer a slightly different perspective on mental wellbeing. A 5-point Likert scale is used, ranging from none of the time (1), to rarely (2), some of the time (3), often (4) and all of the time (5) to indicate the feelings of respondents. The score by summing the scores for all seven items (7-35) before transforming the total score based on the metric score conversion table. Scores range from 7 to 35 and higher scores indicate higher positive mental wellbeing.
Change from Baseline in Risk of Fall Trough Short Falls Efficacy Scale-International (Short FES-I) at 5 weeks. | From enrollment to the end of treatment at 5 weeks
  Measures of "fear of falling" or, more properly, "concerns about falling" among participants. It consists of seven items which measure confidence in performing a range of activities of daily living without falling. A 4-point scale is used ranging from no concern (1) about falling to severe concern (4) about falling. The sum of the items ranges from 7 to 28 with cut-off points of low (7-8), medium (9-13), and high (14-28).
Change from Baseline in Self-efficacy Trough Health beliefs and self-efficacy in exercise questionnaires at 5 weeks. | From enrollment to the end of treatment at 5 weeks
  Reflect the concepts of beliefs about individuals' ability to perform exercise and self-efficacy. It consists of twenty items which are: self-efficacy for exercise (four items), barriers to exercise (three items), benefits of exercise (five items), and impact of exercise on arthritis (eight items). A 5-point Likert scale is used ranging from 'strongly agree' to 'strongly disagree' to indicate the beliefs of respondents. The total score is calculating by adding together the respondents scores on the subscale and the sum of the items indicates higher scores reflecting greater self-efficacy or firmer belief in exercise.
Change from Baseline in Quality of Life Trough Knee Injury and Osteoarthritis Outcome Score (KOOS) subscales of quality of life at 5 weeks. | From enrollment to the end of treatment at 5 weeks
  KOOS subscales of quality of life is specifically focuses on assessing the impact of knee problems on a person's quality of life that includes aspects such as how knee issues affect daily activities, recreational activities, and overall well-being. It consists of four items and every item have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included.
Change from Baseline in Pain Trough 11 Point Numerical Rating Scale (NRS) at 5 weeks. | From enrollment to the end of treatment at 5 weeks
  1. NRS - Zero is equivalent to no pain and 10 indicates the worst possible pain.

IPD SHARING:
Plan to Share IPD: No